CLINICAL TRIAL: NCT02052999
Title: An Open Label Pilot Study to Evaluate the Efficacy of PAC-14028 in the Treatment of Erythematotelangiectatic Rosacea and Papulopustular Rosacea
Brief Title: Study to Evaluate the Efficacy and Safety of PAC-14028 Cream in Rosacea Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRPV1-ROSACEA_IIT
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Erythematotelangiectatic Rosacea; Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — N-(1-(3,5-difluoro-4-methanesulfonylaminophenyl)ethyl)-3-(2-propyl-6-trifluoromethylpyridine-3-yl)acrylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PAC-14028 cream 1% (Experimental): PAC-14028 cream 1%, twice daily for 8 weeks
  Interventions: Drug: PAC-14028 cream 1%
- Rozex gel 0.75% (Active Comparator): Rozex gel 0.75%, twice daily for 8 weeks
  Interventions: Drug: Rozex gel 0.75%
- Vehicle (Placebo Comparator): Vehicle, twice daily for 8 weeks
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: PAC-14028 cream 1% — Participants received topical PAC-14028 cream 1% twice daily for 8 weeks
  Other Names: PAC-14028
  Arms: PAC-14028 cream 1%
Other: Vehicle — Participants received topical Vehicle twice daily for 8 weeks
  Other Names: Vehicle of PAC-14028 Cream
  Arms: Vehicle
Drug: Rozex gel 0.75% — Participants received topical Rozex gel 0.75% twice daily for 8 weeks
  Arms: Rozex gel 0.75%

SUMMARY:
The objective of this study is to determine the efficacy and safety of PAC-14028 1% cream of Amorepacific Corporation in patients with erythema-telangiectatic or papulopustular rosacea

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at the age of 20 to 65 years old
* Clinical diagnosis of erythematotelangiectatic or papulopustular rosacea according to National Rosacea Committee Expert Society with

  * Erythema severity ≥ 1
  * Telangiectasia severity ≥ 1
  * At least 3 papules or pustules in facial region
* IGA score ≥ 2
* Voluntarily signed written informed consent forms for study participation

Exclusion Criteria:

* Patients who are unable to be diagnosed or evaluated for rosacea due to tattoo or scar in the facial area
* Patients who are unable to be diagnosed or evaluated for rosacea due to excess hair(e.g., mustache, beard, whiskers etc.) in the facial area
* Patients who are sensitive to the drug or vehicle
* Previous administration of oral retinoid or vitamin A(≥10,000 units/day) within 6 months prior to visit 1
* Previous use of estrogen or oral contraceptives within 3 months prior to visit 1
* Previous use of topical retinoids or oral antibiotics (e.g., tetracycline, tetracycline derivatives, erythromycin, erythromycin derivatives, sulfamethoxazole, trimethoprim) or oral steroid for the treatment of facial rosacea within 1 month prior to visit 1
* Previous use of topical steroid or topical antibiotics, topical treatment for rosacea(e.g., metronidazole, azelaic acid) within 2 weeks prior to visit 1
* Presently undergoing anti-coagulant therapies
* History of hematologic disease
* Ocular-only, Phymatous rosacea, or papulopustular rosacea patients who require systemic antibiotics
* History of laser treatment for rosacea within 6 weeks prior to visit 1
* Alcoholic or drug abuse patients
* Patients who are treated with prohibited concomitant drugs or considered to inevitably require treatment with prohibited concomitant drugs during the study period
* Renal function impairment with creatinine level higher than twice of maximum normal range
* Hepatic function impairment with AST/ALT higher than twice of maximum normal range
* Pregnant and lactating woman, woman with child-birth potential(should have negative pregnancy test at the baseline visit of the study)
* Participation in another clinical study within 1 month prior to screening
* Patients considered ineligible for study participation by the principal investigator or sub-investigator for other reasons; rosacea due to other medical (liver disease, renal failure, etc.), psychotic, or neuropathic causes rather than as a skin disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Investigator Global Assessment (IGA) | Baseline through Study Week 8

SECONDARY OUTCOMES:
Erythema severity | Baseline through Study Week 8
Telangiectasia severity | Baseline through Study Week 8
Inflammatory lesion counts | Baseline through Study Week 8

CONTACTS AND LOCATIONS:
Overall Officials: BeomJoon Kim, Professor, Principal Investigator — Department of Dermatology, Chungang University Hospital
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea